CLINICAL TRIAL: NCT00645645
Title: Genetic Analysis of Brain Disorders
Brief Title: A Study of the Genetic Analysis of Brain Disorders
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980249; 98-HG-0249; NCT00341978 (obsolete NCT alias)
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Holoprosencephaly
Keywords: Holoprosencephaly; Agenesis of Corpus; Callosum; Genetic Tests
MeSH Terms: conditions — Holoprosencephaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- holoprosencephaly (HPE): individuals with overt or subtle clinical findings consistent with the HPE spectrum are eligible to participate

SUMMARY:
A study of the complex genetics of brain development will be undertaken with an emphasis on those genes that cause the most common structural brain anomaly in humans called holoprosencephaly (HPE). This malformation of the brain can result from either environmental or genetic causes, and it is the aim of these investigations to determine the genes responsible for both normal and abnormal brain development through the study of patients with this disorder. Mutations in one such gene, Sonic Hedgehog, have been shown by us to be responsible for approximately one quarter of familial cases of HPE. Other genes either related to the hedgehog pathway or located at unrelated defined genetic loci may also contribute to HPE and are the subject of active investigation. We anticipate that many genes important for normal brain development will be identified in the search for genetic causes of HPE.

DETAILED DESCRIPTION:
Holoprosencephaly (HPE) covers a nearly continuous spectrum of midline abnormalities ranging from unmistakable cyclopia with absence of forebrain separation to mild microforms, such a single central incisor.

The objective of these studies is to identify genetic factors (coding and non-coding) that contribute to the pathogenesis of holoprosencephaly (HPE) or related brain malformations. Our approach involves common genetic strategies including mutational analysis of candidate genes. All individuals with overt or subtle clinical findings consistent with the HPE spectrum are eligible to participate. Mutational analysis of our entire coded collection of HPE probands (approximately 600 cases) in selected genes is the principal research method used to determine that a given candidate gene is commonly mutated in HPE. This approach pertains to an individual gene(s) or genetic element(s) as well as to targeted capture panels that study gene sets of hundreds of developmental genes whose involvement in brain development is supported by the basic research literature. We are also asking to include the option of investigating the entire set of genetic factors present in the DNA or RNA of patients who have HPE through a proposed change in the consent documents. Whenever a sequence variant is identified, that is not present in a commercially available control set of samples, attempts are made to test the functional significance of this change on the protein itself, or its expression. Sequence changes with a strong probability of being medically significant will be verified in a CLIA-approved lab (e.g. Muneke lab, for selected genes, or commercial lab) at our expense, before any results are given to the family through genetic counseling. Parental DNA (and rarely that of siblings) is usually obtained at the same time that a proband is enrolled. Typically, these samples are studied only to perform limited family studies once a sequence variant of potential medical significance has already been determined. Participation by direct blood relatives is encouraged since virtually all bone fide mutations are either family-specific or de novo. Such family information is critical for the research determination of genetic risk factors and accurate genetic counseling.

The majority of subjects enrolled in this study will continue under the care of their local physician or genetic counselor with limited contact with the NIH investigators. Only rarely will families be seen at the NIH CC. These visits will involve face-to-face genetic counseling of medically significant results, following verification in a CLIA approved lab. This is not a treatment protocol. Our empiric ability to generate medically significant research results is limited by the extensive genetic and other etiologic heterogeneity. Therefore, for most participants this research is not a diagnostic study.

We have modified our procedures to test all new probands for mutations in the four HPE genes (SHH, ZIC2, SIX3 and TGIF). As new genetic elements that confer a risk for HPE are identified, we intend to add additional tests to this panel. Our lab is now certified to receive and test new samples according to CLIA guidelines. However, all previously collected samples will not be considered suitable for diagnostic purposes; hence, a second sample will need to be requested in these cases for CLIA confirmation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. This research is open to all participants with a known or suspected diagnosis of HPE or related brain malformations. Since the range of severity of HPE is extensive, we accept cases compatible with a wide HPE spectrum of findings. All races and genders are known to be at risk for HPE, anywhere in the world. Nationality or place of origin are not specific barriers to participation, provided that a blood tissue sample can be safely sent by international FedEx (to be billed to our account).
  2. Direct blood relatives (typically parents, and occasionally siblings of affected individuals) of patients with HPE are also eligible to participate.
  3. Pregnant women with a fetus with imaging evidence of holoprosencephaly. Most pregnancies affected by holoprosencephaly do not survive to term; therefore, pregnant women will be included in the study. DNA obtained from pregnant women (amniocytes and blood) will be analyzed for genetic etiologies. This will allow for recurrence risk assessment and genetic counseling.

EXCLUSION CRITERIA:

1. Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.
2. Medical condition(s) or cognitive impairment are not in themselves reason for exclusion if in the judgement of the referring physician this would involve no more than minimal risk. We anticipate that children with mental handicaps would be included in the research population. We will make every effort to explain the study for the purpose of assent in a matter that the family feels is both age and developmentally appropriate for that child.
3. We generally review a brief clinical description from the referring physician about a potential research subject to determine that the subject is appropriate to enter into the study. We reserve the right to exclude cases that are clearly not HPE or related to our direct research interests (e.g. HPE cases due to Trisomy 13 or 18 might not be considered directly related to current research). This almost never happens, and we would attempt to make referrals to a more appropriate investigator before a sample is sent to the NIH. Although not desirable, we will accept samples with a suspected diagnosis of HPE where this determination was made by the referring physician independent of any input from our HPE team. In such circumstances, we would likely verify by correspondence that a sample had been received and request further information.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HPE.
Sampling Method: Non-Probability Sample
Enrollment: 5735 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
natural history | lifetime/ongoing
  The objectives of this study are primarily to increase our understanding of the genetic causes of brain malformations.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Solomon, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Belloni E, Muenke M, Roessler E, Traverso G, Siegel-Bartelt J, Frumkin A, Mitchell HF, Donis-Keller H, Helms C, Hing AV, Heng HH, Koop B, Martindale D, Rommens JM, Tsui LC, Scherer SW. Identification of Sonic hedgehog as a candidate gene responsible for holoprosencephaly. Nat Genet. 1996 Nov;14(3):353-6. doi: 10.1038/ng1196-353. PMID 8896571
- [Background] Cohen MM Jr. Perspectives on holoprosencephaly: Part I. Epidemiology, genetics, and syndromology. Teratology. 1989 Sep;40(3):211-35. doi: 10.1002/tera.1420400304. PMID 2688166
- [Background] Cohen MM Jr, Sulik KK. Perspectives on holoprosencephaly: Part II. Central nervous system, craniofacial anatomy, syndrome commentary, diagnostic approach, and experimental studies. J Craniofac Genet Dev Biol. 1992 Oct-Dec;12(4):196-244. PMID 1494025
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1998-HG-0249.html